CLINICAL TRIAL: NCT01155882
Title: Whipple at the Splenic Artery - A Procedure for Ductal Adenocarcinoma of the Pancreas With Extensive Involvement of the Porto-Mesenteric Axis: A Registry Study
Brief Title: Registry Study - Whipple at the Splenic Artery
Acronym: WATSA
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 10-0767 / 201105335
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whipple Surgery at the Splenic Artery: Whipple at the Splenic Artery (WATSA) is at resecting tumors with negative microscopic margins (R0) at the resection line on the pancreas and at the tangential posterior, uncinate, and venous margins.
  Interventions: Procedure: Whipple at the Splenic Artery (WATSA)

INTERVENTIONS:
Procedure: Whipple at the Splenic Artery (WATSA)

SUMMARY:
The purpose of this study is to determine how effective Whipple at the Splenic Artery (WATSA).

DETAILED DESCRIPTION:
Primary

The primary objective of this registry study is to collect clinical data from patients who undergo the WATSA procedure. Specific hypotheses to be tested are

* To determine how effective Whipple at the Splenic Artery (WATSA) is at resecting tumors with negative microscopic margins (R0) at the resection line on the pancreas and at the tangential posterior, uncinate, and venous margins.
* To determine if WATSA can be performed within the usual range of morbidity and mortality (30 day postoperative mortality) for a standard a Whipple procedure.

Secondary

The secondary objectives of this registry study are to

* To determine the survival/recurrence rates at 2 years.
* To determine the effect of occlusion of the splenic vein at the confluence.

ELIGIBILITY:
Eligibility Criteria - Prospective Portion:

* Patient must have diagnosis of ductal adenocarcinoma of head and/or neck of pancreas, ampullary adenocarcinoma, or pancreatic neuroendocrine tumor confirmed by tissue diagnosis.
* Patient must be between 18 to 85 years of age.
* Patient must be a candidate for the WATSA procedure or have had the WATSA surgery performed within 1 year.
* Patient must be able to understand and willing to sign a written informed consent document.

Eligibility Criteria - Retrospective Portion:

Patient underwent WATSA procedure at our institution between 01/01/2009 and 12/31/2011.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from PI's patient population or referrals from colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Effectivity of the Whipple at the Splenic Artery | By CT scan at 8 weeks post surgery
  To determine how effective Whipple at the Splenic Artery (WATSA) is at resecting tumors with negative microscopic margins (R0) at the resection line on the pancreas and at the tangential posterior, uncinate, and venous margins.
To determine range of morbidity and mortality | 30 day postoperative mortality
  To determine if Whipple at the splenic artery can be performed within the usual range of morbidity and mortality (30 day postoperative mortality) for a standard a Whipple procedure.

SECONDARY OUTCOMES:
Survival/recurrence at 2 years | 2 years
  To determine the survival/recurrence rates at 2 years.
Effect of occlusion of the splenic vein at the confluence. | By CT scan at 8 weeks
  To determine the effect of occlusion of the splenic vein at the confluence.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Strasberg, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu